CLINICAL TRIAL: NCT03206775
Title: Collection of Normative Data for iPad-Based Cognitive Assessment Tools
Brief Title: D2D Normative Data for Remote Assessments
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of California, San Francisco (Other); Posit Science Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: STUDY00000319
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Cognition
Keywords: cognitive training; Self-report assessments; Normative Data
MeSH Terms: interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Healthy controls (Phase 1): Participants will participate in Cognitive Assessments (Phase 1) developed by Posit Science
  Interventions: Behavioral: Cognitive Assessments (Phase 1)
- Healthy Controls, Battery A (Phase 2): Participants will complete the Cognitive Battery A (Phase 2) developed by Posit Science while at the Minnesota State Fair.
  Interventions: Behavioral: Cognitive Battery A (Phase 2)
- Healthy Controls, Battery B (Phase 2): Participants will complete the Cognitive Battery B (Phase 2) developed by Posit Science while at the Minnesota State Fair.
  Interventions: Behavioral: Cognitive Battery B (Phase 2)
- Healthy Controls, Battery C (Phase 2): Participants will complete the Cognitive Battery C (Phase 2) developed by Posit Science while at the Minnesota State Fair.
  Interventions: Behavioral: Cognitive Battery C (Phase 2)
- Healthy Controls (Phase 3): Participants will complete the full Posit Science cognitive assessment battery and self-report questionnaires for credit in the Research Experience Program at the University of Minnesota.
- Healthy Controls, Battery D (Phase 2): Participants will complete the Cognitive Battery E (Phase 2) developed by Posit Science while at the Minnesota State Fair.
- Healthy Controls, Battery E (Phase 2): Participants will complete the Cognitive Battery C (Phase 2) developed by Posit Science while at the Minnesota State Fair.
- Adolescents with anxiety diagnosis (Phase 4): Participants will complete remote cognitive assessments and cognitive training programs developed by Posit Science.
- Adolescents, healthy controls (Phase 4): Participants will complete remote cognitive assessments and cognitive training programs developed by Posit Science.

INTERVENTIONS:
Behavioral: Cognitive Assessments (Phase 1) — Participants will participate in up to 6 assessments in 4 domains of cognition: Processing Speed; Executive Attention; Learning and Memory; and Social Cognition.
  Assessments:
  * Visual Sweeps
  * Sustained Visual Attention
  * Associative Learning--Visual
  * Associative Learning--Auditory
  * Emotion Motion
  * Voice Choice
  Groups: Healthy controls (Phase 1)
Behavioral: Cognitive Battery A (Phase 2) — Participants will complete two visual assessments, one auditory assessment, and one social cognition assessment. Then the participant will complete self-report surveys.
  Assessments:
  * On trails: Learning
  * Line Length Discrimination
  * Tap the Emotion
  * Sound Sweeps
  * BIS/BAS
  * TEPS
  * Feasibility survey
  Groups: Healthy Controls, Battery A (Phase 2)
Behavioral: Cognitive Battery B (Phase 2) — Participants will complete two visual assessments, one auditory assessment, and one social cognition assessment. Then the participant will complete the complete self-report surveys.
  Assessments:
  * Visual Time Order Judgment
  * Target Tracker
  * Emotional Face
  * Auditory Sound Discrimination
  * BIS/BAS
  * TEPS
  * Feasiblity assessment
  Groups: Healthy Controls, Battery B (Phase 2)
Behavioral: Cognitive Battery C (Phase 2) — Participants will complete two visual assessments, one auditory assessment, and one social cognition assessment. Then the participant willcomplete self-report surveys.
  Assessments:
  * Stroop 2AFC
  * Visual Task Switcher
  * Beep Seeker
  * Voice Choice
  * BIS/BAS
  * TEPS
  * Feasibility Survey
  Groups: Healthy Controls, Battery C (Phase 2)

SUMMARY:
Phase 1: This is a remote observational study in which participants will complete cognitive assessments developed by Posit Science. Participants will be healthy controls aged 18-65 with reliable internet access and a device that they can use to access the assessments, such as a laptop or iPad. Participants will complete up to 6 Posit Science assessments in different domains of cognition, which should last approximately 30 minutes.

Phase 2: This is an in person observational study in which participants will complete cognitive assessments developed by Posit Science. Participants will be healthy controls aged 18-80 who are fluent in English. Participants will complete batteries of cognitive assessments developed by Posit Science, which include combinations of visual, auditory, and social cognitive assessments, and self-report questionnaires. This study will be conducted at the Driven to Discover building at the Minnesota State Fair. Participation will last approximately 20 minutes.

Phase 3: Participants in Phase 3 will complete a Posit Science assessment battery and self-report questionnaires. Each participant will be asked to provide brief demographic and medical history data. Participants will be aged 18-35 and will be students at the University of Minnesota who are enrolled in the Research Experience Points program. Participants will complete the assessment battery remotely; the battery will take approximately 45-60 minutes to complete.

Phase 4: This is a pilot program to test the use of remote cognitive assessment and training in adolescents with an anxiety diagnosis and healthy controls. Participants will complete a short assessment battery, then will receive 4 hours of cognitive training over 2 weeks at home. Then they will repeat the battery. Total participation should last approximately 5 hours over 2-3 weeks and will be completed entirely remotely.

DETAILED DESCRIPTION:
Phase 1: Remote Assessment with Old Battery (Enrollment period: June-August 2017. CLOSED TO ENROLLMENT) Participants who have successfully completed the online consent process may begin study procedures. A member of the research staff will connect the participant to the Posit Science battery remotely using their laptop or iPad through the BrainHQ portal. All Posit Science assessments have a brief training section before the assessment begins. Participants will be instructed to be in a quiet place free of distractions where they can turn up the volume on their device or use headphones to complete the auditory portions of the assessment. The battery will consist of 6 exercises and will last approximately 20 minutes, which will be completed in a single sitting. Data to be captured will include response time, accuracy, and time to complete the assessment. These data will be stored confidentially within the Posit Science servers and will later be downloaded onto an external device for data analysis and interpretation. Once participants have completed the batter, a member of the study staff will send their compensation.

Phase 2: Minnesota State Fair (Enrollment period: 2017-2022) Participants who have successfully completed the consent process may begin study procedures. A member of the research staff will connect the participant to the REDCap self-report surveys on an iPad. The surveys will be contained within a directory listed under the participant's unique study identifier and will not contain any personally identifying information. The first survey will collect demographic information such as age, gender, ethnicity/race, zip code of residence, education level, current medications, and personal and familial psychiatric and neurological history. This information will be collected in a self-report survey form to avoid embarrassment or stigma that could result if the participant was overheard answering these questions. After completing the demographic survey and brief medical history, all participants will complete self report questionnaires. The self-report assessments should take approximately 2 minutes to complete.

After the completion of the self-report items, the participant will be automatically redirected to the cognitive battery to which they have been randomized. They will be asked to log in to the BrainHQ portal using the same email address they provided before. They will be prompted for their name; study staff will instruct participants to enter "State" for their first name and "Fair" for their last name. However, study staff will not directly oversee participants while they create their account, and so some may not follow these instructions and may disclose their full name to Posit Science. All Posit Science assessments have a brief training section before the assessment begins. If the participant is still having trouble understanding the assessment, study staff will be available to help explain the tasks. Participants will be provided with over-the-ear headphones with disposable sanitary pads for auditory components. Each battery will consist of 4-6 Posit Science assessments, which last approximately 2-3 minutes each. The cognitive battery should last approximately 12-15 minutes. Data to be captured will include response time, accuracy, and time to complete the assessment. These data will be stored confidentially within the Posit Science servers and will later be downloaded onto an AHC managed device for analysis and interpretation. When downloaded to the AHC server, they will be de-identified and collated using a unique participant ID.

At the end of the cognitive assessment battery, participants will be asked to complete a short feasibility survey on REDCap which will ask them their opinion of the tasks they completed and how likely they would be to use these kinds of programs. This survey should take approximately 1-2 minutes. Then participants will receive their compensation and their participation will be complete.

Phase 3: Research Experience Program (REP) Project (Enrollment period: Spring 2018; future enrollment planned) Adult students at the University of Minnesota who are enrolled in the Research Experience Points (REP) program may enroll in this study to be awarded points for class credit. We will request that participants complete the study in a quiet environment free of distractions with a reliable internet connection, and that they do not participate if they have consumed alcohol or illicit substances in the last 8 hours/are under the influence of illicit substances. We will also recommend the use of over-the-ear headphones for the study. Participants will complete an online consent form independently, though they may contact research staff at any time if they have questions. After completing the consent form, participants will be redirected to the COMPAS self-report measures. After the assessment suite is complete, the participants will be automatically re-directed to the Posit Science website to complete the assessment battery. Total participation should take approximately 45-60 minutes.

Phase 4: Pilot Adolescent Cognitive Training (Enrollment period: Summer 2018. CLOSED TO ENROLLMENT) We will recruit adolescents without a mental health diagnosis and with a diagnosis of anxiety by using the UMP Psychiatry Clinic recruitment registry, contacting previous research participants, by advertising in the community and online (Facebook and Department website). Parents/guardians will be asked to provide a brief demographic and medical history about their child. If the participant is over 18, they may complete this independently, but are instructed that they can work with their parent or guardian if they choose to do so. The adolescent will then complete the assessment battery, 4 hours of BrainHQ training games over 2 weeks, and repeat the assessment battery. Total participation should last approximate 5 hours and will be completed entirely remotely. Participants will receive their compensation via email, using the same account that was used for sending the link to the battery

ELIGIBILITY:
Phase 1 Inclusion Criteria:

* Aged 18-65
* Willing and able to provide informed consent as determined by the REDCap assessment
* Fluent in English (learned before the age of 12)
* Has reliable internet access and a device such as a laptop or iPad which can be used to connect to the BrainHQ portal in a quiet place free of distraction
* Able to use an iPad or computer to perform visual and auditory cognitive assessments unassisted
* No history of schizophrenia, bipolar disorder with psychosis, or schizoaffective disorder
* No neurological disorder, major head injury, mental retardation diagnosis, or autism spectrum disorder
* Pregnant women may participate in this study

Phase 2 Inclusion Criteria:

* Aged 18-80
* Willing and able to provide informed consent
* Learned English before the age of 12
* Pregnant women may participate in this study
* Able to use an iPad to perform visual and/or auditory cognitive assessments unassisted.

Phase 3 Inclusion Criteria:

* Aged 18-35
* Willing and able to provide informed consent Fluent in English Able to use an iPad or computer to perform visual and auditory cognitive assessments unassisted
* Has reliable internet access and a device such as a laptop or iPad which can be used to connect to the REDCap server and BrainHQ portal in a quiet place free of distraction

Phase 4 Inclusion Criteria:

* Aged 12-18
* Either has no mental health diagnosis (healthy control) or is diagnosed with an anxiety disorder
* Willing and able to provide assent; at least one parent or guardian is able to provide written consent for participation
* Fluent in English
* Consistent access to a device with the iOS operating system (e.g., iPhone, iPad)
* Able to use an iOS device to perform visual and auditory cognitive assessments unassisted
* Has reliable internet access in a quiet place free from distraction to complete study activities

Exclusion Criteria for all participants:

* Unable or unwilling to provide informed consent
* Not fluent in written/spoken English
* Unable to use an iPad or computer to complete visual and/or auditory cognitive assessments without assistance
* Presence of a medical or behavioral condition that would prohibit participation in the trial
* Participant has used illicit substances or alcohol within the past 8 hours

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Phase 1: Participants in this study will be healthy adults, aged 18-65, who are fluent in English and do not have a history of schizophrenia, schizoaffective disorder, bipolar disorder with psychotic features, autism spectrum disorder, mental retardation, neurological disorder, or history of major head injury. Participants will not be restricted by their geological location as they can access the study portal remotely with a reliable internet connection. Pregnant women may participate in this study.
  Phase 2: Participants in this study will be attendants of the Minnesota State Fair, aged 18-80, who learned English before the age of 12 and can use an iPad without assistance. Participants may be pregnant or have a medical, developmental, psychiatric, or neurological condition.
Sampling Method: Non-Probability Sample
Enrollment: 1271 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Visual Sweeps | 4 minutes
  Phase 1: Participants watch two spatial frequency sweeps and determine whether each one swept inward or outward
Sustained Visual Attention | 4 minutes
  Phase 1: Participants are asked to press the spacebar as fast as they can whenever a star appears at the top of the screen (don't press when it appears at the bottom of the screen)
Associative Learning--Visual | 4 minutes
  Phase 1: Participants will see a ring of items. They are asked to memorize the items and their locations.
Associative Learning--Auditory | 4 minutes
  Phase 1: Participants will hear a sequence of syllables. They are asked to memorize the syllables and repeat the sequence by clicking on the words.
Emotion Motion | 4 Minutes
  Phase 1: Participants will see a video of a person showing a facial expression on every trial. They are asked to select the correct emotion
Voice Choice | 4 Minutes
  Phase 1: A sentence spoken in a certain prosody will be presented on every trial. Correctly choose the emotion expressed in the sentence
On Trails: Learning | 4 minutes
  Phase 2, Battery A: Participants see two circles connected by paths. Remember the path from A to B, and click the circles in the order indicated. If the participant makes a mistake, the path is shown again.
Line Length Discrimination | 4 minutes
  Phase 2, Battery A: Participants watch two lines surrounded by stars and determine which one is longer.
Tap the Emotion | 4 minutes
  Phase 2, Battery A: This is an executive function go/no-go task that captures both inhibitory control and sustained attention abilities. Participants see a series of faces, each presented for a limited time. Participants are instructed to tap the button every time they see a happy or sad face, and to not tap the button when they see a neutral face
Sound Sweeps | 4 minutes
  Phase 2, Battery A: Participants are presented with two subsequent tones that eithe rrise or lower in pitch, and they are asked to identify the direction of the pitch change.
Visual Time Order Judgment | 4 minutes
  Phase 2, Battery B: Watch two visual patterns shown one after the other and determine which one was presented first
Target Tracker | 4 minutes
  Phase 2, Battery B: Keep track of the targets as all the objects (targets and distractors) move around the screen.
Emotional Face | 4 minutes
  Phase 2, Battery B: This is an emotional stroop task that provides a measure of executive attention. In each trial, an expressive face is shown and overlaid with a congruent or incongruent word (stroop effect). Participants see a series of faces, each presented for a limited time. Identify the emotion of the face as quickly as possible. If the face is displaying happiness, tap the HAPPY button. If the face is displaying fear, tap the FEAR button. Increased reaction time to incongruent stimulus combinations capture capacity for conflict resolution.
Auditory Sound Discrimination | 4 minutes
  Phase 2, Battery B: Participants must determine which of two similar sounding syllable phonemes were spoken.
Stroop 2AFC | 4 minutes
  Phase 2, Battery C: The name of a color written in colored text appears in the screen. Participants elect the color of the text by tapping left/right keyboard arrow as quickly as they can.
Visual Task Switcher | 4 minutes
  Phase 2, Battery C: Two shapes are presented rapidly on the screen. Respond quickly if the two shapes share the same criteria, which changes from trial to trial (e.g., color).
Beep Seeker | 4 minutes
  Phase 2, Battery C: Participants are presented with a target beep tone and then asked to identify it in the presence of distracting tones.
Voice Choice | 4 minutes
  Phase 2, Battery C: A sentence spoken in a certain prosody will be presented on every trial. Correctly choose the emotion expressed in the sentence

SECONDARY OUTCOMES:
Behavioral Inhibition Scale/Behavioral Activation Scale (BIS/BAS) | 4 minutes
  Participants will answer self-report questions to determine behavioral inhibition and behavioral activation. The scale is set at 1-4 1 not active at all and 5 being the most active
Temporal Experience of Pleasure Scale (TEPS) | 4 minutes
  Participants will answer self-report questions to determine their anticipatory and consummatory pleasure. Scale range is 1-6 1 being least pleasurable and 6 being the most pleasurable
Feasibility ratings | 1 minute
  Participants will answer self report questions about the accessibility of the Posit Science cognitive assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - University of Minnesota, Dept of Psychiatry, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided